CLINICAL TRIAL: NCT06311786
Title: A Phase 1, Open-Label Study to Investigate the Absorption, Distribution, Metabolism, and Excretion of Single Oral Dose [14C]-BIIB091 in Healthy Male Participants
Brief Title: A Study to Look at How a Single Oral Dose of Carbon-14-Labelled [14C] BIIB091 Moves Through and is Processed by the Body in Healthy Male Participants
Acronym: Mass Balance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 257HV107
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-BIIB091 (Experimental): Participants will receive a single oral dose of [14C]-BIIB091 on Day 1.
  Interventions: Drug: [14C]-BIIB091

INTERVENTIONS:
Drug: [14C]-BIIB091 — Administered as specified in the treatment arm.

SUMMARY:
The main goal of this study is to learn how [14C]-BIIB091 moves through and is processed by the body and to look at how much of BIIB091's metabolites (what is produced when BIIB091 is broken down by the body) appears in the blood, urine, and stool in healthy male participants. The study will also help researchers learn more about the safety of BIIB091 in healthy male participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index (BMI) of 18 to 32 kilograms per meter square (kg/m^2) and a total body weight greater than (>) 50 kg, as measured at Screening.
* History of regular bowel movements (averaging 1 or more bowel movements per day).
* Negative polymerase chain reaction (PCR) test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Day -1.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease or other major disease, as determined by the Investigator.
* Participants enrolled in a previous radionucleotide study within 12 months prior to screening or who have received radiotherapy within 12 months prior to screening or such that total radioactivity would exceed acceptable dosimetry.
* Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia), as determined by the Investigator, within 90 days prior to Screening or between Screening and Day -1.
* Current enrollment in any other drug, biological, device, or clinical study or treatment with an investigational drug or approved therapy for investigational use within 30 days prior to Day -1 (24 weeks for biologics), or 5 half-lives, whichever is longer.
* Prior exposure to BIIB091 or any lymphocyte-depleting therapy or exposure to any lymphocyte-targeting therapy within 3 months prior to Day -1.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Amount of BIIB091 Excreted per Sampling Interval in Urine (Aeu) | Pre-dose and at multiple timepoints up to Day 10
Amount of BIIB091 Excreted per Sampling Interval in Feces (Aef) | Pre-dose and at multiple timepoints up to Day 10
Cumulative Amount of BIIB091 Excreted per Sampling Interval in Urine (Cum Aeu) | Pre-dose and at multiple timepoints up to Day 10
Cumulative Amount of BIIB091 Excreted per Sampling Interval in Feces (Cum Aef) | Pre-dose and at multiple timepoints up to Day 10
Percentage of BIIB091 Excreted per Sampling Interval in Urine (%Feu) | Pre-dose and at multiple timepoints up to Day 10
Percentage of BIIB091 Excreted per Sampling Interval in Feces (%Fef) | Pre-dose and at multiple timepoints up to Day 10
Cumulative Percentage of BIIB091 Excreted in Urine (Cum %Feu) | Pre-dose and at multiple timepoints up to Day 10
Cumulative Percentage of BIIB091 Excreted in Feces (Cum %Fef) | Pre-dose and at multiple timepoints up to Day 10
Maximum Observed Concentration (Cmax) of [14C]-BIIB091-Derived Materials in Plasma and Whole Blood | Pre-dose and at multiple timepoints up to Day 5
Time to Reach Maximum Observed Concentration (Tmax) of [14C]-BIIB091-Derived Materials in Plasma and Whole Blood | Pre-dose and at multiple timepoints up to Day 5
Area Under the Concentration-Time Curve From Time 0 to Time of the Last Measurable Concentration (AUClast) of [14C]-BIIB091-Derived Materials in Plasma and Whole Blood | Pre-dose and at multiple timepoints up to Day 5
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of [14C]-BIIB091-Derived Materials in Plasma and Whole Blood | Pre-dose and at multiple timepoints up to Day 5
Terminal Half-Life (t1/2) of [14C]-BIIB091-Derived Materials in Plasma and Whole Blood | Pre-dose and at multiple timepoints up to Day 5
Apparent Clearance (CL/F) of BIIB091 in Plasma | Pre-dose and at multiple timepoints up to Day 5
Apparent Volume of Distribution (Vz/F) of BIIB091 in Plasma | Pre-dose and at multiple timepoints up to Day 5
Quantitative Profile of [14C]-BIIB091 Metabolites in Plasma | Pre-dose and at multiple timepoints up to Day 4
Quantitative Profile of [14C]-BIIB091 Metabolites in Urine | Pre-dose and at multiple timepoints up to Day 10
Quantitative Profile of [14C]-BIIB091 Metabolites in Feces | Pre-dose and at multiple timepoints up to Day 10

SECONDARY OUTCOMES:
Cmax of Plasma Metabolite 23 (M23) | Pre-dose and at multiple timepoints up to Day 5
Tmax of Plasma M23 | Pre-dose and at multiple timepoints up to Day 5
AUClast of Plasma M23 | Pre-dose and at multiple timepoints up to Day 5
AUCinf of Plasma M23 | Pre-dose and at multiple timepoints up to Day 5
t1/2 of Plasma M23 | Pre-dose and at multiple timepoints up to Day 5
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to end of study follow-up (Day 11)
Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Parameters | From Day 1 up to Day 10
Number of Participants With Clinically Significant Vital Sign Abnormalities | From Day 1 up to Day 10
Number of Participants With Clinically Significant Physical Examination Abnormalities | From Day 1 up to Day 10
Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities as Assessed by 12-Lead ECG Measurements | From Day 1 up to Day 5
Number of Participants With Change in Columbia Suicide Severity Rating Scale (C-SSRS) Score | From Day 1 up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- PPD Clinical Research Unit, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/